CLINICAL TRIAL: NCT01642667
Title: The Efficacy and Safety of Pharmacoinvasive Therapy With Prourokinase for Acute ST Segment Elevation Myocardial Infarction Patients With Expected Percutaneous Coronary Intervention Related Delay
Brief Title: Pharmacoinvasive Therapy With Prourokinase
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Landing Pharmaceuticals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PROUK
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — saruplase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- primary PCI (Placebo Comparator)
  Interventions: Drug: Placebo
- prouk-PCI (Active Comparator)
  Interventions: Drug: Prourokinase

INTERVENTIONS:
Drug: Prourokinase — a bolus of 1.2 million IU and an infusion of 4.8 million IU in 60 min.
  Arms: prouk-PCI
Drug: Placebo
  Arms: primary PCI

SUMMARY:
The aim of this study is to elucidate the efficacy and safety of pharmacoinvasive therapy by using prourokinase (prouk), a unique fibrin-specific agent, in patients with ST-segment elevation myocardial infarction (STEMI)

ELIGIBILITY:
Inclusion Criteria:

* age 75 years or younger, symptom onset 6 h or less before randomization, intention to undertake primary PCI, ST-segment elevation of 2 mm or more in two anterior leads or of 1 mm or more in two inferior leads if they had ST-segment elevation, or new left bundle-branch block.

Exclusion Criteria:

* expected arrival at the catheterization laboratory less than 1 h or more than 3 h after randomization, anticipated problems with vascular access, previous enrollment to other studies, and the usual contraindications to thrombolytic therapy.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
angiographic parameters which can demonstrate the myocardium reperfusion, including TIMI flow grade (grade I-III), TIMI frame count (frame) and myocardial blush grade (MBG,grade 0-3). | 90 minutes after prourokinase bolus

SECONDARY OUTCOMES:
major adverse cardiac events [MACE, defined as the composite of all cause-death, reinfarction, revascularization (including target vessel and non-target vessel revascularizations), or rehospitalization due to new or worsening congestive heart failure] | 12 month after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Shenyang Northern Hospital, Shenyang, Liaoning, China

REFERENCES:
- [Derived] Han YL, Liu JN, Jing QM, Ma YY, Jiang TM, Pu K, Zhao RP, Zhao X, Liu HW, Xu K, Wang G, Wang B, Sun RH, Wang J. The efficacy and safety of pharmacoinvasive therapy with prourokinase for acute ST-segment elevation myocardial infarction patients with expected long percutaneous coronary intervention-related delay. Cardiovasc Ther. 2013 Oct;31(5):285-90. doi: 10.1111/1755-5922.12020. PMID 23634911